CLINICAL TRIAL: NCT04356560
Title: SARS-CoV-2 Surveillance of Patients and Healthcare Workers at the Department of Otorhinolaryngology, Head and Neck Surgery and Audiology, Rigshospitalet University Hospital of Copenhagen, Denmark
Brief Title: COVID-19 Surveillance of Patients and Healthcare Workers in a Hospital Department
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ramon Gordon Jensen, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: DT P-2020-353
Record Dates: First submitted 2020-04-13; First posted 2020-04-22 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: healthcare worker; infection control; otorhinolaryngology; epidemiology
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — oropharyngeal swabs, nasopharyngeal swabs, blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthcare workers: Actively working at Department of Otorhinolaryngology Head and Neck Surgery & Audiology, Rigshospitalet University Hospital of Copenhagen, Denmark. During 2020 COVID 19 pandemic
  Interventions: Diagnostic Test: COVID-19 test, polymerase chain reaction for SARS-CoV-2
- Patients: Patients presenting with complications to upper respiratory tract infections and patients undergoing surgery involving airway mucosa During 2020 COVID 19 pandemic
  Interventions: Diagnostic Test: COVID-19 test, polymerase chain reaction for SARS-CoV-2

INTERVENTIONS:
Diagnostic Test: COVID-19 test, polymerase chain reaction for SARS-CoV-2 — surveillance
  Other Names: COVID-19 blood samples, immunoglobuline levels

SUMMARY:
Doctors, nurses and staff members of ear-nose and throat (ENT) departments are at high risk due to aerosol-inducing diagnostic procedures and surgery during the COVID-19 epidemic. Reports from China, Spain, Italy and England report of fatal cases among ENT specialists. With a concurrent lack of personal protection, it is of paramount importance to identify patients and healthcare workers at an early stage to prevent a COVID-19 outbreak in the department. A baseline study of all healthcare workers has been performed. Follow-up will be accomplished by interval testing, antibody measurements and REDcap Covid-19 questionnaires. All patients at risk of carrying SARS-CoV-2, or who are candidates for high-risk airway surgery will be tested. Infection control measures at the department will be implemented progressively according to the real-time surveillance results from both patients and healthcare workers.

DETAILED DESCRIPTION:
At present the COVID-19 pandemic is evolving, and numbers of cases admitted to hospital and case fatalities are on the rise in Denmark.

The epidemic of SARS-CoV-2 can pose a great burden on all healthcare systems at both national and local level.Data from the SARS epidemic (2002-2003) showed that the countries with the largest number of cases were China (including administrative regions), Canada and Singapore.Healthcare workers accounted for 20%,43% and 41%, respectively of the total number of cases.

In the initial stages of the current pandemic, Wuhan ear-nose and throat (ENT) doctors were affected at higher rates than other doctors at the hospital (personal message from Stanford University, confirmed in media). This has been acknowledged by the Confederation of European Otorhinolaryngology - Head and Neck Surgery (CEORL HNS). A possible explanation is the close contact with the patient's airway mucosa during routine ENT examinations, the risk of inducing sneezing and coughing during these examinations and the use of nasal endoscopic procedures among other airway procedures,at both examination and during surgery. Compared to SARS, the new SARS-CoV-2 seems to have a higher viral load in the nasopharynx, posing increased risk for ENT doctors.

Persons who experience symptoms from the airways are in Denmark advised to stay at home, as they may have COVID-19, and only contact the health care system if the situation deteriorates. However, unspecific symptoms or complications in the upper airways, the oral cavity, pharynx and neck can lead to contact with an ENT department, e.g. in case of symptoms potentially related to cancer. Bacterial super infections as complications to viral airway infections is seen during e.g. influenza epidemics. Acute bacterial middle ear infections is one of the most common infections among children and is associated with virus in 80 % of cases. Complications include acute mastoiditis, ethmoiditis and peritonsillar abscess,which are potentially life-threatening conditions which need to be treated at a hospital ENT department. It is not known if the incidence of these bacterial super infections will increase during the SARS-CoV-2 pandemic or if such an increase will lead to a concurrent increase in the exposure of virus to the healthcare workers within the ENT departments.

COVID-19 has a broad spectrum of clinical presentations from asymptomatic, to complicated pneumonias, to multi-organ failure and death. Studies have shown that 2/3 of patients with SARS-CoV-2 will have debut of symptoms from the upper airways.

Protecting and monitoring healthcare workers and patients The mode of human transmission for SARS-Cov-2 is not fully understood, but expected to be through direct contact and partly by aerosol transmission, which is the reason for the health authorities' current advice of keeping distance.

SARS-Cov-2 can remain viable as aerosols for more than three hours, with a half-life of 1.1 hours and on plastic surfaces for up to 72 hours with a half-life of 6.8 hours.

Virus has shown to be present in the oropharynx the first week after symptom onset with a subsequent decline, but viral RNA has been detected up to 25 days after.

The use of personal protection including mask and gloves are essential for healthcare workers treating patients with COVID-19.

However, on March 3rd 2020 The World Health Organization announced global shortage of personal protection supplies. In Denmark, there is also a current shortage of adequate protection, which increases the risk for healthcare workers as the epidemic intensifies in the population.

Large scale population testing in Iceland indicates that half of individuals carrying SARS-CoV-2 are asymptomatic. With a concurrent lack of personal protection in a department with a high risk of SARS-CoV-2 exposure, it is important to identify infected patients and infected healthcare workers at an early stage,in order to prevent a COVID-19 outbreak within the department.

As the Danish healthcare system was not prepared for an epidemic of this nature, detailed guidelines to reduce transmission to healthcare workers at department level are deficient. The department will progressively implement infection disease control measures based on monitored real time data from the patient and healthcare worker surveillance. Control measures will follow local guidelines and be inspired by recommendations from departments who managed the SARS epidemic.

ELIGIBILITY:
Inclusion Criteria:

1. Healthcare workers of all professions with daily routines at the Department of Otorhinolaryngology Head and Neck Surgery & Audiology, Rigshospitalet University Hospital of Copenhagen
2. All patients with symptoms of upper respiratory tract infections
3. All patients undergoing surgery involving the mucosa of the upper airways

Exclusion Criteria:

1. healthcare workers not affiliated to the department
2. Patients without symptoms of upper respiratory tract infection (e.g otitis externa, fractures)
3. Patients undergoing surgery not involving the upper airway (e.g thyroidectomy, Neck)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Danish healthcare workers. variation in socioeconomic background. Majority lives in Greater Copenhagen area
  2. Danish patients all ages, variation in socioeconomic background. Patients with cancers tends to be older, higher prevalence of comorbidities. Live in eastern region of Denmark. Patients with upper airway complications to infections tend to be younger and without comorbidities. Majority from Greater Copenhagen area
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of healthcare workers with SARS-CoV-2 | 6 months
  Change from baseline in number of healthcare workers positive for SARS-CoV-2. Measured by repetitive naso/oropharyngeal swab tests of all active healthcare workers at the department.
Incidence of ENT patients with SARS-CoV-2 | 6 months
  Change from baseline in number of patients positive for SARS-CoV-2. Measured by naso/oropharyngeal swab tests
Development of SARS-CoV-2 antibodies among healthcare workers | 6 months
  Incidence and prevalence of SARS-CoV-2 antibodies by repetitive blood samples testing SARS-CoV-2 antibody levels of immunoglobulin G and immunoglobulin M

SECONDARY OUTCOMES:
Sensitivity and specificity of a COVID-19 screening symptom questionnaire among healthcare workers | 6 months
  Compare number of positive questionnaires with number of positive oro/nasopharyngeal swab test and antibody tests
SARS CoV-2 and bacterial super infections in upper respiratory airways | 6 months
  Change from baseline in total number of complications to upper respiratory tract infections (URTI). Proportion of SARS CoV-2 positives among patients with URTI compared to proportion of SARS CoV-2 positive among ENT patients with non-infectious disease (eg cancer)

CONTACTS AND LOCATIONS:
Overall Officials: Inge J Knudsen, MD, Study Chair — Rigshospitalet, Department of Microbiology; Nikolai S Kirkeby, MSc, Study Chair — Rigshospitalet, Department of Microbiology; Ramon G Jensen, MD, Principal Investigator — Rigshospitalet, Dep. of ORL, Head and neck & Audiology
Locations (1):
- Rigshospitalet University Hospital of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Individual anonymized participant data can be made available on request